CLINICAL TRIAL: NCT00231777
Title: A Randomized, Double-Blind, Active Comparator-Controlled, Parallel-Group Study Conducted Under In-House Blinding Conditions, to Examine the Safety and Tolerability of IV MK0517 for the Prevention of Postoperative Nausea and Vomiting (PONV)
Brief Title: A Study to Examine the Safety and Tolerability of MK0517 for the Prevention of Post-Operative Nausea and Vomiting (0517-015)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0517-015; 2005_074
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2010-06-08 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Post-Operative Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 40 mg MK0517 IV
  Interventions: Drug: Comparator: MK0517
- 2 (Active Comparator): 4 mg ondansetron IV
  Interventions: Drug: Comparator: ondansetron

INTERVENTIONS:
Drug: Comparator: MK0517 — a single administration of 40 mg MK0517 by IV immediately prior to surgery
  Arms: 1
Drug: Comparator: ondansetron — a single administration of 4 mg ondansetron by IV immediately prior to surgery
  Other Names: Zofran
  Arms: 2

SUMMARY:
A new intravenous medication is being tested for the prevention of the nausea and vomiting that occurs after surgery. This new medication is being compared to another intravenous medication that is already available to patients for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Open abdominal surgery requiring 24 hour hospital stay
* General anesthesia
* Post-operative opioids
* ASA status of I-III

Exclusion Criteria:

* Patient exhibits evidence of any clinically significant respiratory, metabolic, hepatic, renal dysfunction, or cardiovascular condition or congestive heart failure (CHF)
* Morbid obesity
* Patient is mentally incapacitated or has a significant emotional or psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2005-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 02-Aug-2005; Last Patient Out: 29-Nov-2005; 15 study centers in the US
Pre-assignment Details: Patient is at least 18 years of age and is scheduled to undergo open abdominal surgery or vaginal hysterectomy requiring overnight hospital stay (24-hour hospital stay after end of surgery).
Groups:
- MK0517 Intravenous (IV) 40 mg: On Day 1-All patients assigned to the MK0517 treatment group were administered 1 vial of MK0517 40 mg and 1 vial of matching sterile normal saline 0.9% placebo for ondansetron.
- Ondansetron IV 4 mg: On Day 1- All patients assigned to the ondansetron treatment group were administered 1 vial of ondansetron 4 mg and 1 vial of matching sterile normal saline 0.9% placebo for MK0517.
Period: Overall Study
Arm/Group | MK0517 Intravenous (IV) 40 mg | Ondansetron IV 4 mg
Started | 170 | 46
Completed | 164 | 44
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- MK0517 Intravenous (IV) 40 mg: On Day 1-All patients assigned to the MK0517 treatment group were administered 1 vial of MK0517 40 mg and 1 vial of matching sterile normal saline 0.9% placebo for ondansetron.
  Data Reported is for all all participants who received active study therapy.
- Ondansetron IV 4 mg: On Day 1- All patients assigned to the ondansetron treatment group were administered 1 vial of ondansetron 4 mg and 1 vial of matching sterile normal saline 0.9% placebo for MK0517.
  The formulation of MK0517 used in this study was a non polysorbate (PS80) formulation which was not further developed and is not available for use.
  Data Reported is for all all participants who received active study therapy.
- Total: Total of all reporting groups
Arm/Group | MK0517 Intravenous (IV) 40 mg | Ondansetron IV 4 mg | Total
Number analyzed (Participants) | 167 | 44 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.01) | 43.3 (8.51) | 45.8 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 42 | 203
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5 | 1 | 6
  Black | 20 | 7 | 27
  Hispanic American | 17 | 5 | 22
  Native American | 1 | 0 | 1
  White | 124 | 31 | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs)
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: Baseline and 24 hours
Population: All patients as treated (APaT) which included all patients who received active study therapy.
Measure: Number; unit: Participants
Arm/Group | MK0517 Intravenous (IV) 40 mg | Ondansetron IV 4 mg
Number analyzed (Participants) | 167 | 44
Participants | 125 | 32

2. Primary Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs)
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product.
Time Frame: Baseline and 24 hours
Population: All patients as treated (APaT) which included all patients who received active study therapy.
  patients in the MK0517 40 mg treatment group were randomized but did not have at least one post-baseline laboratory test and therefore were not counted as part of the N analyzed.
Measure: Number; unit: Participants
Arm/Group | MK0517 Intravenous (IV) 40 mg | Ondansetron IV 4 mg
Number analyzed (Participants) | 165 | 44
Participants | 9 | 2

3. Secondary Outcome: Number of Patients With Drug-related CAEs
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs
Time Frame: Baseline and 24 hours
Population: All patients as treated (APaT) which included all patients who received active study therapy.
Measure: Number; unit: Participants
Arm/Group | MK0517 Intravenous (IV) 40 mg | Ondansetron IV 4 mg
Number analyzed (Participants) | 167 | 44
Participants | 33 | 8

4. Secondary Outcome: Number of Patients With Serious CAEs
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: Baseline and 24 hours
Population: All patients as treated (APaT) which included all patients who received active study therapy.
Measure: Number; unit: Participants
Arm/Group | MK0517 Intravenous (IV) 40 mg | Ondansetron IV 4 mg
Number analyzed (Participants) | 167 | 44
Participants | 15 | 3

ADVERSE EVENTS:
Time Frame: 1-day plus 14 days post-therapy
Description: Number of subjects at risk includes randomized subjects who had follow-up and completed the trial after at least one dose of treatment.
Arm/Group | MK0517 Intravenous (IV) 40 mg | Ondansetron IV 4 mg
Serious Adverse Events (participants affected / at risk) | 15/167 | 3/44
Other Adverse Events (participants affected / at risk) | 124/167 | 31/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0517 Intravenous (IV) 40 mg (N=167) | Ondansetron IV 4 mg (N=44)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pelvic Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Bladder Injury (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Anoxic Encephalopathy (Nervous system disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Pelvic Congestion (Reproductive system and breast disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal Laceration (Reproductive system and breast disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0517 Intravenous (IV) 40 mg (N=167) | Ondansetron IV 4 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 12 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 7 | 2
Extrasystoles (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 6 | 0
Eye Irritation (Eye disorders) | 1 | 0
Eye Pain (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 18 | 8
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 7 | 0
Flatulence (Gastrointestinal disorders) | 12 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 47 | 12
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2
Chest Pain (General disorders) | 2 | 0
Chills (General disorders) | 4 | 2
Fatigue (General disorders) | 1 | 0
Feeling Jittery (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Infusion Site Erythema (General disorders) | 7 | 0
Infusion Site Induration (General disorders) | 9 | 0
Infusion Site Oedema (General disorders) | 1 | 0
Infusion Site Pain (General disorders) | 18 | 3
Infusion Site Reaction (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 5 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 12 | 3
Cellulitis (Infections and infestations) | 1 | 0
Fungal Rash (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 3
Vaginal Infection (Infections and infestations) | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1
Delayed Recovery From Anaesthesia (Injury, poisoning and procedural complications) | 1 | 0
Suture Rupture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion Reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Body Temperature Increased (Investigations) | 0 | 1
Oxygen Saturation Decreased (Investigations) | 0 | 1
Urine Output Decreased (Investigations) | 5 | 0
Calcium Deficiency (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 18 | 8
Migraine (Nervous system disorders) | 2 | 0
Neuropathy (Nervous system disorders) | 0 | 1
Paraesthesia Oral (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 14 | 5
Restlessness (Psychiatric disorders) | 0 | 1
Bladder Perforation (Renal and urinary disorders) | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Oliguria (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 8 | 4
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Vulval Laceration (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 10
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticari (Skin and subcutaneous tissue disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 11 | 0
Hypotension (Vascular disorders) | 16 | 7
Phlebitis (Vascular disorders) | 5 | 0

LIMITATIONS AND CAVEATS:
The formulation of MK0517 used in this study was a non polysorbate (PS80) formulation which was not further developed and is not available for use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.